CLINICAL TRIAL: NCT03704623
Title: Parecoxib vs Paracetamol in the Treatment of Acute Renal Colic Due to Ureteric Calculi: Randomized Controlled Trial
Brief Title: Parecoxib vs Paracetamol in the Treatment of Acute Renal Colic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: Amiri Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Professor of Urology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Parecoxib vs Paracetamol
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Acute Renal Colic; Ureteric Stone
Keywords: Acute renal colic; Ureteric stone; Selective COX2 inhibitor; Parecoxib; Paracetamol
MeSH Terms: conditions — Renal Colic; Ureterolithiasis | interventions — Acetaminophen; parecoxib

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to one of the two treatment groups.
Who Masked: Participant, Investigator
Masking Description: The emergency department (ED) nurse will do randomization by drawing one of the sealed closed envelopes that contain the analgesic to be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Active Comparator): Patients will receive IV 1 g of Paracetamol
  Interventions: Drug: Paracetamol
- Parecoxib (Active Comparator): Patients will receive 40 mg of Parecoxib IV
  Interventions: Drug: Parecoxib

INTERVENTIONS:
Drug: Paracetamol — Paracetamol 1g IV
  Other Names: Perfalgan
  Arms: Paracetamol
Drug: Parecoxib — Parecoxib 40 mg IV
  Other Names: Dynastat
  Arms: Parecoxib

SUMMARY:
This study will be conducted to compare the efficacy and safety of Parecoxib versus Paracetamol for treatment of acute renal colic due to ureteric stones.

DETAILED DESCRIPTION:
Eligible patients will be randomized to one of the two treatment groups. Group 1 patients will receive IV 1 g of Paracetamol while group 2 patients will receive 40 mg of Parecoxib IV.

The Visual Analogue Scale (VAS) will be calculated on presentation and at 30 minutes after analgesia administration. Patients who do not respond to an initial dose of the analgesia will receive rescue analgesia in the form of Morphine, 01.mg/kg, IV.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms consistent with acute renal colic

Exclusion Criteria:

* Hypersensitivity to either Paracetamol or Parecoxib.
* History of peptic ulcer.
* Pregnant or breastfeeding females.
* Patients with hepatic impairment (Child-Pugh score >10).
* Patients with chronic kidney disease (CKD) Stage 4 or 5 (eGFR <30mls/min).
* History of coronary ischemia, peripheral vascular or cerebrovascular disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
The need for rescue analgesia (Morphine) | 30 minutes
  Patient who had persistent pain

SECONDARY OUTCOMES:
The incidence of adverse effects due to medication used | 24 hours
  Assessment of adverse effects of the drug used

CONTACTS AND LOCATIONS:
Overall Officials: Abdullatif AL-Terki, MD, Study Chair — Amiri Hospital
Locations (1):
- Al-Amiri Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No